CLINICAL TRIAL: NCT05848037
Title: Assessment of CymActive™ Catheter Technology for UrinAry ReTention and AcceptancE (The ACCTUATE Study)
Acronym: ACCTUATE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow study recruitment within the current protocol and the time required to implement an amended study protocol led the Sponsor decision to cease participant recruitment and to discontinue the study.
Sponsor: Ingenion Medical Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MF2208-A-R0001
Record Dates: First submitted 2023-04-24; First posted 2023-05-08 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-06

CONDITIONS: Urinary Retention
Keywords: Urinary retention; Catheter; urology; urinary catheter; Quality of Life; TURP; Trans Urethral Resection of the Prostate; Randomised Controlled Study; RCT; CAUTI; Catheter Associated Urinary Tract Infection; novel; new; magnet; valve; patient
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Intervention Model Description: Two treatment arms with patients randomised 1:1, into treatment arm (cymactive™ catheter) and routine standard of care arm (Foley-type catheter).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cymactive™ catheter device (CCD) arm (Experimental): Approximately 60 participants will be recruited to this study. Approximately 30 patients in the CCD arm.
  Interventions: Device: cymactive™ catheter device (CCD)
- Foley-type device (FTD) arm (Active Comparator): Approximately 60 participants will be recruited to this study. Approximately 30 patients in the FTD treatment group.
  Interventions: Device: Foley-type catheter device

INTERVENTIONS:
Device: cymactive™ catheter device (CCD) — The cymactive™ catheter (manufactured by Ingenion Medical Ltd) received CE marking on the 28th March 2024, as a Class IIb device (n. ECM24MDR002 rev.0, Single Registration Number (SRN) of the Manufacturer UK-MF-000041065) and will be available in the UK market, subject to local arrangements.
  The cymactive™ catheter is designed to remain in situ for up to 30 days, does not extend outside the patient's body except for 2 removal strings, and has an integral, magnetically controlled valve that allows the user to control their own urination. The study participant will each be supplied with a magnetic Actuator (a separate Class I device supplied by Ingenion Medical) so they are in control of valve and their own voiding. The magnet is strong and care will need to be taken to keep it at least 6 inches from magnetically-sensitive items, i.e. mobile phones, laptops and credit cards. Study participants should also avoid contact with MRI machines.
  Arms: cymactive™ catheter device (CCD) arm
Device: Foley-type catheter device — Routine standard of care. Usually replaced ~ 3 monthly
  Arms: Foley-type device (FTD) arm

SUMMARY:
The ACCTUATE study: Assessment of CymActive™ Catheter Technology for UrinAry reTention and acceptancE study will evaluate a novel catheter design that addresses the specific needs of male long term catheter users living in the community. The primary endpoint of the study will be tolerability, assessed by measuring patient-reported Quality of Life and VAS pain scale assessments up to approximately day 90 (end of study). The secondary endpoints will be comparisons of the Adverse Event nature and frequency, up to approximately 90 days (end of study) and genomic profiling of the abundance and diversity of microorganisms present in the screening visit urine sample versus the end of study urine sample of participants from both arms of the trial.

DETAILED DESCRIPTION:
There is an urgent need to address sub-optimal catheterisation that some men experience when living in the community with urinary retention problems. The catheters currently used within the NHS and in community settings are typically of the Intermittent or 'Foley' type. Foley type catheters are based on a nearly 100-year-old design, where an inflatable balloon, filled with water which anchors one end of the catheter within the bladder. At the other end, external to the body, a bag collects the urine, or a valve allows its discharge. Another option for patients requiring catheters is intermittent self-catheterisation. Intermittent catheters are single use, and self-catheterisation is needed multiple times per day, in order to empty the bladder. The number of times an intermittent catheter is used depends on the patient's condition and the frequency is guided by a Health Care Professional.

It is accepted that catheters in their current form, create a burden on the NHS, as Catheter Associated Urinary Tract Infections (CAUTI's) are one of the leading causes of healthcare-associated infections (HCAIs) and contribute significantly to mortality rates. Of Foley-type and intermittent users, the Foley- type catheters tend to lead to more infections.

The cymactive™ catheter (manufactured by Ingenion Medical Ltd) received CE marking on the 28th March 2024, as a Class IIb device (n. ECM24MDR002 rev.0, Single Registration Number (SRN) of the Manufacturer UK-MF-000041065). The cymactive™ catheter is designed to remain in situ for up to 30 days and does not extend outside the patient's body, except for two removal strings. The catheter has an integral, magnetically controlled valve that allows the user to control their own urination.

Study participants will be supplied with a magnetic Actuator (a separate Class I device supplied by Ingenion Medical), so they are in control of the valve and their own voiding.

The manufacturers of the cymactive™ catheter anticipate that the device may result in a better patient experience and potentially, a reduced risk of CAUTI when compared to a Foley catheter.

ACCTUATE is a multi-centre study, comparing the cymactive™ catheter device (CCD) versus Foley-type devices (FTD) in men with non-neurogenic urinary retention.

Study participants will be randomised (1:1) to receive either the cymactive™ catheter or a Foley catheter (the control arm) and the relevant catheter will be inserted on day 1 of the study. The cymactive™ catheters will be replaced approximately every 30 days, with a total study duration of approximately 90 days. Study participants randomised to the Active Comparator arm will receive the standard of care catheter (Foley) on day 1, for approximately 90 days. At the end of study visit (approx. day 90), CCD-treated subjects will undergo the removal of the CCD and a return to standard of care treatment, typically a FTD. However, as the cymactive™ device is CE marked, there is the possibility that the device may be available for post-study use, dependent upon clinical opinion and cymactive™ availability at specific institutions.

Approximately 60 participants will be recruited to this study; 30 patients in the CCD arm and 30 patients in the FTD arm.

The study will begin with the recruitment of a Sentinel group of 20 patients consisting of 10 patients randomised to the CCD arm and 10 patients randomised to the FTD arm. A review of the Sentinel group data, up to day 30 of the study, may be undertaken to examine any potential futility and/or safety signals. The Sentinel group will continue to participate in the study during this time as detailed in the Schedule of Activities.

Participants will be male adults (≥ 18 years) with a documented history of non-neurogenic urinary retention and long-term catheter use (> or = 4 weeks).

ELIGIBILITY:
Inclusion Criteria:

Participants will be eligible to enrol in the study only if all of the following apply

* Male (anatomical)
* Adult, more than or equal to 18 years of age
* Capacity to give written informed consent
* Documented urinary retention, this may include patients who await a TURP, or similar, procedure
* Non-neurogenic urinary retention
* Catheter use on a long-term basis (>4 weeks)

Exclusion Criteria:

Participants will not be eligible to enrol in the study if any of the following apply

* Symptomatic bacteriuria (at screening)
* Surgical procedures performed in the lower urinary tract
* Neurogenic urinary retention
* Patients who have had a TURP (or similar) procedure
* Any malignancy in active/radical treatment (note: subjects with prostate or bladder cancer under surveillance only, may be enrolled into the study, at the Investigator's discretion)
* Patients who have a pacemaker or significant cardiovascular disease
* Participants with any contraindications, as outlined in the IFU
* Active participation in another interventional trial within the last 30 days
* Any condition, abnormality or issue, for which the investigator assesses the subject as unsuitable for an interventional study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The device is designed for use in individuals who have a urethral length of between 11 - 16cm. As such, the device is not able to treat women or other people with a urethral length that is less than 11cm. The study will only recruit anatomically male subjects.
Enrollment: 6 (Actual)
Dates: Start 2025-05-29 (Actual); Primary Completion 2025-10-10 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
To evaluate tolerability of the cymactive™ catheter device (CCD) compared to Foley-type devices (FTD) as assessed by patient-reported Quality of Life questionnaire. | Up to approximately 90 days
  Tolerability will be assessed using the validated Quality of Life questionnaire (ICIQ-LTCqol). The intervention cymactive™ catheter arm will be compared against the control, Foley type device, treatment arm.
1. To evaluate tolerability of the cymactive™ catheter device (CCD) compared to Foley-type devices (FTD) as assessed by patient-reported VAS pain scale. | Up to approximately 90 days
  Tolerability will be assessed using VAS pain scale assessments. The intervention cymactive™ catheter arm will be compared against the control, Foley type device, treatment arm.

SECONDARY OUTCOMES:
Comparison of the genomic profile (abundance and diversity) of microorganisms present in the screening visit urine sample versus the end of study urine sample of participants from both arms of the trial. | Up to approximately 90 days
  Genomic profiling of the diversity and abundance of microorganisms providing insight in the microbial populations in the screening and end of study urine samples will be compared for each subject and for each treatment arm in a descriptive way.
1. To evaluate the safety of the cymactive™ catheter device (CCD) compared to Foley-type devices (FTD) as assessed by the nature and frequency of adverse events up to approximately day 90. | Up to approximately 90 days
  All AEs including CAUTIs in both treatment arms will be collected up to approximately study day 90. The proportion of patients with one or more AEs at 90 days and the proportion of patients with one or more CAUTIs will be compared between the CCD and the FTD group using a binomial test.

CONTACTS AND LOCATIONS:
Overall Officials: Hashim Hashim, MBBS, FEBU, FRCS, Principal Investigator — North Bristol NHS Trust; Edward C Cappabianca, BA, MBA, Study Director — Ingenion Medical Ltd.
Locations (5):
- United Kingdom (5):
  - Addenbrookes Hospital - Cambridge University Hospitals NHS Foundation Trust, Cambridge, Cambridgeshire
  - Royal Devon & Exeter Hospital - Royal Devon University Healthcare NHS Trust, Exeter, Devon
  - Ipswich Hospital - East Suffolk and North Essex NHS Foundation Trust, Ipswich, Essex
  - Frimley Park Hospital - Frimley Health NHS Foundation Trust, Camberley, Surrey
  - Southmead Hospital - North Bristol NHS Trust,, Bristol

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Ingenion Medical Ltd Homepage — https://www.ingenionmedical.co.uk
- See also: Urology News Article — https://cloud.3dissue.net/30176/30072/30344/88513/index.html?UROMA23=&utm_source=MA23+Edition&utm_medium=Email&utm_campaign=MA23+Urology+News/?page=23